CLINICAL TRIAL: NCT05434845
Title: The Effect of Blood on the Protein to Creatine Ratio During Pregnancy
Brief Title: The Effect of Blood on the PC Ratio During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marshall University (Other)
Collaborators: University at Buffalo (Other)
Responsible Party: Principal Investigator, Jesse Cottrell, Assistant Professor, Marshall University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1912480
Record Dates: First submitted 2022-06-21; First posted 2022-06-28 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Proteinuria in Pregnancy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Divide urine into 4 different specimen cups with 20 mLs of urine each to measure urinalysis (UA) and PC ratio:
  1. UA and PC ratio on original sample
  2. UA and PC ratio with 1 mL of whole blood added
  3. UA and PC ratio with 2 mL of whole blood added
  4. UA and PC ratio with 5 mL of whole blood added
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- UA and PC ratio on original sample (No Intervention): Original urine sample
- UA and PC ratio with 1 mL of whole blood added (Active Comparator): 1 mL of whole blood added to 20 mLs of urine
  Interventions: Other: Blood draw
- UA and PC ratio with 2 mL of whole blood added (Active Comparator): 2 mL of whole blood added to 20 mLs of urine
  Interventions: Other: Blood draw
- UA and PC ratio with 5 mL of whole blood added (Active Comparator): 5 mL of whole blood added to 20 mLs of urine
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — An additional 8 mL of blood will be drawn during routine lab collection
  Arms: UA and PC ratio with 1 mL of whole blood added; UA and PC ratio with 2 mL of whole blood added; UA and PC ratio with 5 mL of whole blood added

SUMMARY:
This study will examine the effect if blood on the the protein to creatine (PC) ratio in pregnant patients by adding blood to urine samples.

DETAILED DESCRIPTION:
The Purpose of the Research:

The purpose of this study is to examine the effect of blood on the protein to creatine (PC) ratio in pregnant patients.

The Scientific or Scholarly Rationale:

The PC ratio is used to diagnosis proteinuria in pregnancy. It is thought that blood in the urine will cause the PC ratio to be elevated but there are no current studies to prove this hypothesis.

The Procedures to be Performed:

Upon presentation to the Labor and Delivery Triage or the Antepartum Unit, patients will be enrolled in the study. Urine collection that is not needed for medical workup will be collected and saved, and an extra 8 mLs of blood will be drawn during routine lab collection by phlebotomy team. Additional lab costs will be covered by Marshall Obstetrics & Gynecology.

Lab protocol: Divide urine into 4 different specimen cups with 20 mLs of urine each to measure urinalysis (UA) and PC ratio:

1. UA and PC ratio on original sample
2. UA and PC ratio with 1 mL of whole blood added
3. UA and PC ratio with 2 mL of whole blood added
4. UA and PC ratio with 5 mL of whole blood added

Subjects medical records will be reviewed for past obstetrical history after consent to be in the study.

The Risks and Potential Benefits of the Research:

Risks: 8 mLs of additional maternal blood will be drawn for study purposes. Possible risks could include pain, bleeding, fainting, bruising, infection, or hematoma (blood clot under the skin) at the injection site. Please note that routine blood would be drawn regardless of study enrollment.

Benefits: Our hypothesis is that the PC ratio will be elevated by contamination with blood. It is unknown if this hypothesis is correct.

Complete Inclusion/Exclusion Criteria (may be submitted separately if extensive):

Inclusion criteria includes patients presenting to Labor and Delivery Triage or Antepartum Unit at Cabell Huntington Hospital between the ages of 18 and approximately 45 years and gestational age of >20 weeks.

Exclusion criteria includes pre-existing proteinuria (excess protein in the urine) or hematuria (blood in the urine).

ELIGIBILITY:
Inclusion Criteria:

* Labor and Delivery Triage or Antepartum Unit at Cabell Huntington Hospital between the ages of 18 and approximately 45 years and gestational age of >20 weeks

Exclusion Criteria:

* pre-existing proteinuria (excess protein in the urine) or hematuria (blood in the urine)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 20 (Estimated)
Dates: Start 2022-06-19 (Actual); Primary Completion 2022-12-19 (Estimated); Study Completion 2022-12-19 (Estimated)

PRIMARY OUTCOMES:
To measure the PC ratio after whole blood has been serially added | 6 months
  The PC ratio is used to diagnose proteinuria in pregnancy. Our goal is to determine if blood causes the PC ratio to be elevated.

CONTACTS AND LOCATIONS:
Locations (1):
- Marshall University School of Medicine, Huntington, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be accessed by the IRB approved research team